CLINICAL TRIAL: NCT00533000
Title: Short Term Perioperative Smoking Cessation and the Effect on Postoperative Complications. A Randomized Clinical Trial.
Brief Title: Smoking Cessation and Postoperative Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-214
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2007-09

CONDITIONS: Postoperative Complications; Randomized; Prevention; Smoking Cessation
MeSH Terms: conditions — Postoperative Complications; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Smoking cessation
  Interventions: Procedure: Smoking cessation
- B (No Intervention)

INTERVENTIONS:
Procedure: Smoking cessation — Weekly smoking cessation by professional counseling and nicotine substitute on request
  Arms: A

SUMMARY:
The primary aim of this study is to evaluate the effect of preoperative smoking cessation on postoperative complications among patients undergoing surgery. Secondary aims are to evaluate effect on wound complications, short and long term effects including abstinence rate, pain, quality of life and effects on the immune system.

DETAILED DESCRIPTION:
Tobacco smokers suffers from postoperative complications after surgery more extensively than non-smokers. Our primary aim is to study if smoking cessation four weeks prior to elective surgery decreases the number of postoperative complications. Secondary aims is to analyse if smoking cessation four weeks prior to elective surgery decreases wound complications, analyse the effect on abstinence rate, effect on postoperative pain, quality of life and if smoking cessation normalises; the immunological response to surgery.

The study is randomised, prospective, multicenter-based trial. Daily smokers are randomised to 1. Control group (standard care) or 2. smoking cessation. Patients randomised to smoking cessation will undergo professional motivational counselling and will receive free nicotine substitution. The study will include elective cases that are scheduled for surgery. Cessation starts 3-5 weeks prior to surgery. All patients are prospectively followed up for four weeks concerning post-operative complications and for one year concerning other outcomes. Outcome (complications) is registered by a blind observer.

Analyses will be performed by intention to treat. The intervention group is compared with the control group and an adjustment for possible confounders will be done. There will also be an analysis in the subgroups depending on which surgical procedure was performed.Secondary analyses will be by protocol

ELIGIBILITY:
Inclusion Criteria:

* Active, daily tobacco smokers (> 2 cigarettes daily for at least one year prior to inclusion), 18-79 years old at the time of randomisation.
* Proficiency in the Swedish language.
* Oral and written consent.
* Scheduled for primary inguinal hernia repair or other umbilical hernia repair or laparoscopic cholecystectomy
* Scheduled for hip- or knee replacement

Exclusion Criteria:

* - Active drug abuse or severe mental illness prohibiting compliance with the study protocol.
* Pregnancy.
* Residence outside the county of Stockholm.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2004-01; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of any postoperative complication | 1 month

SECONDARY OUTCOMES:
wound complication rate, smoking cessation rates, level of postoperative pain, quality of life, thioredoxin reductase, Il-1, Il-6, TNFa | 1-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Adami, MD, Principal Investigator — Karolinska Institutet

REFERENCES:
- [Derived] Lindstrom D, Sadr Azodi O, Wladis A, Tonnesen H, Linder S, Nasell H, Ponzer S, Adami J. Effects of a perioperative smoking cessation intervention on postoperative complications: a randomized trial. Ann Surg. 2008 Nov;248(5):739-45. doi: 10.1097/SLA.0b013e3181889d0d. PMID 18948800